CLINICAL TRIAL: NCT06308965
Title: Does Vessel-sparing Surgery in Anterior Approach Total Hip Arthroplasty Change Clinical Outcome?
Acronym: USP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z-2023088
Record Dates: First submitted 2024-02-21; First posted 2024-03-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Tensor Fasciae Latae Syndrome; Arthroplasty Complications
Keywords: Total Hip Arthroplasty; Ultra Sparing Procedure; Direct Anterior Approach

STUDY DESIGN:
Intervention Model Description: This is a monocentric prospective randomized blinded clinical trial during a period of minimal 3 years or until 150% of sample size is included (100 patients).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be blinded and randomized into two cohorts. The selection and randomization protocol is as follows: participants eligible for the study are requested to participate and informed by the study nurse. If the patient agreed to participate, informed consent is obtained, and the patient is included in the study. At that time, the study nurse uses a mobile randomization application (Random, Dublin, Ireland) to allocate them either to the 'standard' (sacrificing the vessels) or 'vessel sparing' DAA.
  Weighted randomization (1:2) is applied to compensate for a dropout of patients planned for vessel sparing surgery, but in whom the vessels were damaged unintendedly. In case a bilateral procedure will be performed, each side is randomized individually.
  Surgery will be performed by the surgeon. Data collection before and after surgery is collected by personal assistant who is unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacrificing vessels (Active Comparator)
  Interventions: Procedure: Vessel ligation technique
- Sparing vessels (Experimental)
  Interventions: Procedure: Vessel sparing technique

INTERVENTIONS:
Procedure: Vessel sparing technique — Vessel sparing
  Arms: Sparing vessels
Procedure: Vessel ligation technique — Vessel ligation
  Arms: Sacrificing vessels

SUMMARY:
During direct anterior approach (DAA) for total hip arthroplasty (THA), ligation of the lateral femoral circumflex artery and vessel is always conducted. However, this standardized procedure may jeopardize blood muscle perfusion and cause tenderness in the tensor fascia lata muscle. The investigators want to investigate whether blood vessel-sparing surgery is feasible, reproducible, and would alter outcomes following DAA THA.

The surgical technique of the vessel-sparing procedure will be described and investigated in a prospective blinded RCT. The investigators hypothesize that the vessel-sparing technique is feasible in 60% of the patients. If these vessels were not sacrificed, the investigators expect the incidence of TFL tendinopathy to be lower.

DETAILED DESCRIPTION:
Primary objective: to compare a group with successful vessel-sparing with a vessel-sacrificed-group for:

1. Incidence of TFL tendinopathy
2. Patient-reported outcomes
3. Component placement Secondary objective: to observe the feasibility of the vessel-sparing surgical technique.

This is a monocentric prospective randomized blinded clinical trial during a period of minimum 3 years or until 150% of the sample size is included (100 patients).

ELIGIBILITY:
Inclusion criteria To be eligible to participate in this study, a subject must meet all criteria below;

* Scheduled for THA by Dr. Frans-Jozef Vandeputte or Professor Dr. Kristoff Corten
* Provide signed and dated informed consent
* Males or females age > 18 years

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Neurological problems with sensorial and/or motoric disturbances (Multiple Sclerosis, Parkinson's disease, hemiplegia, …)
* Previous surgery of the ipsilateral hip
* Ipsilateral neck of femur fracture
* Previous contralateral THA
* Significant hip deformity: Crowe type 3 and 4 dysplasia, Leg-Calvé-Perthes
* Avascular necrosis of the femoral head
* Participating in another study that may interfere with participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
a) Incidence of TFL tendinopathy | one year follow-up
  Clinical examination to detect TFL tendinopathy
b-1) Patient-reported outcome 1: modified Harris Hip Score (HHS) | one year follow-up
  modified Harris Hip Score (HHS) minimum (worse) score = 0 maximum (best) score = 44
b-2) Patient-reported outcome 2: Hip And Groin Outcome Score (HAGOS) | one year follow-up
  Hip And Groin Outcome Score (HAGOS) minimum (worse) score = 0 maximum (best) score = 100
b-3) Patient-reported outcome 3: Forgotten Joint Score | one year follow-up
  Forgotten Joint Score minimum (worse) score = 0 maximum (best) score = 100
b-4) Patient-reported outcome 4: Hip disability and Osteoarthritis Outcome Score (HOOS). | one year follow-up
  Hip disability and Osteoarthritis Outcome Score (HOOS) minimum (worse) score = 0 maximum (best) score = 100
c) Component placement (x-rays) | one year follow-up
  Using pelvic anteroposterior radiographs, with both legs internally rotated 15°:
  Acetabular version (Lewinnek method). Acetabular inclination Femoral alignment Under-sizing in case the femoral component is not touching cortical bone.

SECONDARY OUTCOMES:
Vessel sparing succesfull | end of surgery
  Successful Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No